CLINICAL TRIAL: NCT03507400
Title: Treatment of Migraine With Introvision, a Method of Mental Self-regulation - IntroMig: Randomised Waiting-list Control Study
Brief Title: Introvision for Migraine and Headaches
Acronym: IntroMig
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Collaborators: University of Hamburg-Eppendorf (Other); Introvision e.V (Unknown)
Responsible Party: Principal Investigator, Dr. Monika Empl, Principal Investigator, Ludwig-Maximilians - University of Munich
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: IntroMig 632-15
Record Dates: First submitted 2018-03-05; First posted 2018-04-25 (Actual); Results first posted 2025-04-18 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-03

CONDITIONS: Migraine; Chronic Migraine
Keywords: Introvision: mental and emotional self-regulation technique; Mindfulness, perception technique; Migraine
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Intervention Model Description: waiting list control study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- non-waiting list group (Experimental): Intervention: Introvision: mental and emotional self-regulation
  Interventions: Behavioral: Introvision: mental and emotional self-regulation
- waiting list group (Experimental): Intervention: Introvision: mental and emotional self-regulation
  Introvision is teached to participants of the waiting-list group at least 6 weaks or more after first group
  Interventions: Behavioral: Introvision: mental and emotional self-regulation

INTERVENTIONS:
Behavioral: Introvision: mental and emotional self-regulation — Participants learn Introvision

SUMMARY:
To evaluate the effect of Introvision, a mental and emotional self-regulation-technique developed by Angelika C. Wager, as migraine preventative compared to a waiting list group.

DETAILED DESCRIPTION:
Randomized, single-center, waiting-list control group study: Introvision as preventative in Migraine

Randomized, single center, waiting-list group control study to evaluate the effect of Introvison, a mental and emotional self regulation method to reduce headache days in patients with migraine, migraine and tension type headache and chronic migraine. The number of headache days 3 months after completion of the last session of Introvision will be compared with the number of headache days of the waiting list group in the month before the course to learn Introvision.

ELIGIBILITY:
Inclusion Criteria:

* Episodic migraine with at least 5 headache days per month, episodic migraine and tension type headache with at least 5 migraine headache days per month, chronic migraine
* Stable prophylactic headache medication
* Stable non-medication headache prophylaxis (sports, relaxation techniques, …)
* Informed consent

Exclusion Criteria:

* Other causes of headache, symptomatic headaches
* Other primary headaches such as Cluster headache, trigeminal neuralgia, idiopathic facial pain, new daily persistent headache
* Severe depression (more than 13 points in the Beck Depression inventory fast screen (BDI-FS)
* Drug - or alcohol abuse
* Non-compliance, especially significant missing entries in the headache diaries
* Active psychosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2017-09-20 (Actual); Primary Completion 2019-09-11 (Actual); Study Completion 2020-07-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Monika Empl, MD, Principal Investigator — Department of Neurology, Marchioninistr. 15, 81377 Munich, Germany
Locations (1):
- Hospital of the Ludwig-Maximilians-University, Munich, Bavaria, Germany

REFERENCES:
- [Derived] Empl M, Loser S, Spille P, Rozwadowska A, Ruscheweyh R, Straube A. Effects of Introvision, a self-regulation method with a mindfulness-based perception technique in migraine prevention: a monocentric randomized waiting-list controlled study (IntroMig Study). J Headache Pain. 2023 Nov 3;24(1):146. doi: 10.1186/s10194-023-01684-0. PMID 37924063

RESULTS

PARTICIPANT FLOW:
Groups:
- Waiting List Group: Intervention: Introvision: mental and emotional self-regulation
  Introvision is teached to participants of the waiting-list group at least 6 weaks or more after first group
  Introvision: mental and emotional self-regulation: Participants learn Introvision
Period: Overall Study
Arm/Group | Non-waiting List Group | Waiting List Group
Started | 35 | 37
Completed | 22 | 29
Not Completed | 13 | 8
Not completed — discontinued | 5 | 1
Not completed — Lost to Follow-up | 8 | 6
Not completed — Protocol Violation | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Non-waiting List Group | Waiting List Group | Total
Number analyzed (Participants) | 35 | 37 | 72
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.3 (12.0) | 41.5 (10.7) | 42.9 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 32 | 67
  Male | 0 | 5 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 35 | 37 | 72
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Germany | 35 | 37 | 72

OUTCOME MEASURES:

1. Primary Outcome: Number of Headache Days Per Month
Description: The number of headache days per month 3 months after completion of the last session of Introvision will be compared with the number of headache days of the waiting list group in the month before the course to learn Introvision.
Time Frame: approximately 4 months, as the course to learn Introvision and the three individual sessions will take nearly 2 months to be completed, and headaches per month will be assessed in the month 3 months after the last session of Introvision.
Measure: Mean (Standard Deviation); unit: days per month
Arm/Group | Non-waiting List Group | Waiting List Group
Number analyzed (Participants) | 22 | 29
days per month | 10.6 (7.7) | 10.9 (6.3)
Statistical Analysis 1: Comparison: Non-waiting List Group vs Waiting List Group; Test type: Superiority; p = 0.63, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Non-waiting List Group vs Waiting List Group; pooled comparison of the participants of the non-waiting list and the waiting list before and after Introvision; Test type: Superiority; p = 0.003, Wilcoxon (Mann-Whitney); Wilcoxon paired test

2. Secondary Outcome: Headache Intensity
Description: Headache intensity rated by the patients themselves with a scale in the headache diary: weak (=1) , moderate (=2), severe (=3) headache. Scores may range from 1 to 3. Average headache intensity of the attacks per months will be compared three months after the last session of Introvision compared to the values before Introvison.
Time Frame: approximately 5 - 6 months, baseline before introvision training and 3 three months after the last introvision session
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Before Introvision: Intervention: Introvision: mental and emotional self-regulation
  Introvision: mental and emotional self-regulation: Participants learn Introvision
- After Introvision: Intervention: Introvision: mental and emotional self-regulation
  Introvision is teached to participants of the waiting-list group at least 6 weaks or more after first group
  Introvision: mental and emotional self-regulation: Participants learn Introvision
Arm/Group | Before Introvision | After Introvision
Number analyzed (Participants) | 49 | 49
units on a scale | 2.0 (0.5) | 2.0 (0.5)

3. Secondary Outcome: Acute Medication Per Month
Description: The number of days with acute medication against migraine attacks/headache per month 3 months after completion of the last session of Introvision will be compared with the number of days with acute medication per month before Introvision.
Time Frame: approximately 5 - 6 months, baseline before introvision training and 3 three months after the last introvision session
Measure: Mean (Standard Deviation); unit: days per month
Arm/Group | Before Introvision | After Introvision
Number analyzed (Participants) | 47 | 47
days per month | 6.3 (3.6) | 5.0 (3.7)
Statistical Analysis 1: Comparison: Before Introvision vs After Introvision; Test type: Superiority; p = 0.004, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Number of Headache Days Per Month in Pooled Groups Analysis Before and 3 Months After Introvision as Parameter for the Efficacy of Introvision
Description: number of headache days per months in pooled groups analysis before and 3 months after Introvision, measured with the number of headache days per months as in the primary outcome measure, but both groups together compared before Introvision and three months after the last session
Time Frame: approximately 5-6 months
Measure: Mean (Standard Deviation); unit: days per month
Arm/Group | Before Introvision | After Introvision
Number analyzed (Participants) | 49 | 49
days per month | 11.7 (6.5) | 9.8 (7.0)
Statistical Analysis 1: Comparison: Before Introvision vs After Introvision; Test type: Superiority; p = 0.003, Wilcoxon (Mann-Whitney); Wilcoxon paired test

5. Secondary Outcome: Headache Management Self-efficacy Scale-German-short Form (HMSE-G-SF)
Description: The headache specific self-efficacy scale (Headache Management Self-efficacy Scale-German-short form: HMSE-G-SF) consists of 6 items with a 7-point response scale which ranges from 1 (strongly disagree) to 7 (strongly agree).The 6 items measure self-efficacy beliefs, for instance: "There are things I can do to alleviate the headache". The scores for each of the six items are combined to compute the total score, that may range from 6 to 42 points. A higher score indicates a stronger self-efficacy in headache management. It is measured before Introvision and three month after the last session of Introvision.
Time Frame: approximately 5 - 6 months, baseline before introvision training and 3 three months after the last introvision session
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Before Introvision | After Introvision
Number analyzed (Participants) | 46 | 46
score on a scale | 21.7 (7.7) | 26.2 (6.0)
Statistical Analysis 1: Comparison: Before Introvision vs After Introvision; Test type: Superiority; p = 0.001, Wilcoxon (Mann-Whitney); Wilcoxon paired test

6. Secondary Outcome: Headache-Impact Test 6, HIT-6
Description: Impact of headache (Headache-Impact Test 6, HIT-6), compared three months after the last session of Introvision to before introvision. The total score may range from 6 to 78 points, a higher score indicates a higher impact of headaches on daily activities.
Time Frame: approximately 5 - 6 months, baseline before introvision training and 3 three months after the last introvision session
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Before Introvision | After Introvision
Number analyzed (Participants) | 47 | 47
score on a scale | 64.3 (4.2) | 61.4 (5.9)
Statistical Analysis 1: Comparison: Before Introvision vs After Introvision; Test type: Superiority; p = 0.001, Wilcoxon (Mann-Whitney); Wilcoxon paired test

7. Secondary Outcome: Overall Satisfaction of Patients
Description: Patients will be asked whether they would recommend Introvision for headache patients and can choose between "yes" or "no". The number of patients responding "yes" is reported.
Time Frame: approximately 5 - 6 months, baseline before introvision training and 3 three months after the last introvision session
Population: 97% of participants recommended Introvision for migraine patients.
Measure: Count of Participants; unit: Participants
Arm/Group | After Introvision
Number analyzed (Participants) | 46
Participants | 45

8. Other Pre Specified Outcome: Influence of Frequency of Exercises as Exploratory Outcome Measure
Description: Influence of frequency of self-regulation exercises per week on outcome, measured with reduction of headache days per month before and after Introvision.
  The frequency of self-regulation exercises is documented by the patients themselves on average in a month in the headache diary, with a three categories scale: 0 exercise per week; 1-3 exercises per week, more than 4 exercises per week.
Time Frame: approximately 5-6 months
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Patients' Mastery of Introvision as Exploratory Outcome Measure
Description: investigators' estimation of patients' mastery of introvision,. Evaluated by the investigator after the last session in a three category scale: good mastery, moderate mastery, insufficient mastery.
  Does the mastery of introvision influence the reduction of headache days per month?
Time Frame: approximately 5-6 months
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Influence of Side of Headache on Outcome as Exploratory Outcome Measure
Description: Do patients with a predominantly left-sided headache show a greater reduction of headache days per month 3 months after completion of the last session of Introvision compared to patients with predominantely right-sided headache?
Time Frame: approximately 5-6 months
Population: Headache days before and after Introvision in patients with a) predominantly left-sided headache, b) predominantly right-sided headache, c) bilateral or equally alterating headache
Measure: Mean (Standard Deviation); unit: days per month
Groups:
- Patients With Predominantly Left-sided Headache Before Introvision: Patients with headache predominantly (estimated more than 70%) on the left side before introvision
- Patients With Predominantly Left-sided Headache After Introvision: Patients with headache predominantly (estimated more than 70%) on the left side after introvision
- Patients With Predominantly Right-sided Headache Before Introvision: Patients with headache predominantly (estimated more than 70%) on the right side before introvision
- Patients With Predominantly Right-sided Headache After Introvision: Patients with headache predominantly (estimated more than 70%) on the right side after introvision
- Patients With Bilateral or Alternating Headache Before Introvision: Patients with bilateral headache or headaches that alternate both sides equally before introvison
- Patients With Bilateral or Alternating Headaches After Introvision: Patients with bilateral headache or headaches that alternate both sides equally after introvison
Arm/Group | Patients With Predominantly Left-sided Headache Before Introvision | Patients With Predominantly Left-sided Headache After Introvision | Patients With Predominantly Right-sided Headache Before Introvision | Patients With Predominantly Right-sided Headache After Introvision | Patients With Bilateral or Alternating Headache Before Introvision | Patients With Bilateral or Alternating Headaches After Introvision
Number analyzed (Participants) | 12 | 12 | 16 | 16 | 23 | 23
days per month | 13.9 (5.7) | 10.1 (3.6) | 9.9 (4.5) | 9.1 (4.9) | 11.7 (7.3) | 10.4 (9.4)
Statistical Analysis 1: Comparison: Patients With Predominantly Left-sided Headache Before Introvision vs Patients With Predominantly Left-sided Headache After Introvision; Test type: Superiority — Wilcoxon paired test; p = 0.04, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Patients With Predominantly Right-sided Headache Before Introvision vs Patients With Predominantly Right-sided Headache After Introvision; Test type: Superiority; p = 0.25, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Patients With Bilateral or Alternating Headache Before Introvision vs Patients With Bilateral or Alternating Headaches After Introvision; Test type: Superiority; p = 0.02, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: Start of group sessions till forth month after last introvision session, when collecting the data after the last Introvision session (diaries, questionnaires, question for recommendations) participants were asked whether they experienced any adverse events.
Groups:
- Introvision Group: Intervention: Introvision: mental and emotional self-regulation
  Introvision: mental and emotional self-regulation: Participants learn Introvision
- Waiting List Group Before Introvision: Intervention: Introvision: mental and emotional self-regulation
  Introvision is teached to participants of the waiting-list group at least 6 weaks or more after first group
  Introvision: mental and emotional self-regulation: Participants learn Introvision
Arm/Group | Introvision Group | Waiting List Group Before Introvision
All-Cause Mortality (participants affected / at risk) | 0/51 | 0/37
Serious Adverse Events (participants affected / at risk) | 0/51 | 0/37
Other Adverse Events (participants affected / at risk) | 1/51 | 0/37
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Introvision Group (N=51) | Waiting List Group Before Introvision (N=37)
Tachycardia self-limiting during a SAP (stating attentive perception) exercise (Cardiac disorders) | 1 (1) | 0 (0) — after Introvision training

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (6):
  • Study Protocol: Cover letter EC (2015-10-22): https://cdn.clinicaltrials.gov/large-docs/00/NCT03507400/Prot_003.pdf
  • Study Protocol: EC application (2015-10-22): https://cdn.clinicaltrials.gov/large-docs/00/NCT03507400/Prot_004.pdf
  • Study Protocol: EC Form (2015-10-22): https://cdn.clinicaltrials.gov/large-docs/00/NCT03507400/Prot_005.pdf
  • Study Protocol: Study Protocol without Cover letter wo Application wo Form (2025-03-30): https://cdn.clinicaltrials.gov/large-docs/00/NCT03507400/Prot_006.pdf
  • Statistical Analysis Plan (2015-10-13): https://cdn.clinicaltrials.gov/large-docs/00/NCT03507400/SAP_002.pdf
  • Informed Consent Form (2025-03-30): https://cdn.clinicaltrials.gov/large-docs/00/NCT03507400/ICF_007.pdf